CLINICAL TRIAL: NCT05652894
Title: A Randomized Phase III Study of HX008 (a Humanized Monoclonal Antibody Against PD-1) Compared to Investigator's Choice Chemotherapy in the First-Line Treatment of Subjects With Microsatellite Instability-High (MSI-H)/Deficient DNA Mismatch Repair (dMMR) Metastatic Colorectal Cancer
Brief Title: A Study of HX008 Compared to Chemotherapy in the First-Line Treatment of Subjects With MSI-H/dMMR Metastatic Colorectal Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Taizhou Hanzhong biomedical co. LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HX008-III-CRC-01
Record Dates: First submitted 2022-11-26; First posted 2022-12-15 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Colorectal Neoplasms Intestinal Neoplasms Bevacizumab Cetuximab Irinotecan Oxaliplatin Antibodies Antibodies Monoclonal Antine
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HX008 (Experimental): Subjects receive HX008 200 mg intravenous (IV) every 3 weeks (Q3W)
  Interventions: Drug: HX008
- Investigator's Choice Chemotherapy (Active Comparator): 1. mFOLFOX6
  2. mFOLFOX6+Bevacizumab
  3. mFOLFOX6+Cetuximab
  4. FOLFORI
  5. FOLFORI+Bevacizumab
  6. FOLFORI+Cetuximab
  Interventions: Drug: Investigator's Choice Chemotherapy

INTERVENTIONS:
Drug: HX008 — Drug: HX008 200 mg ,Q3W
  Arms: HX008
Drug: Investigator's Choice Chemotherapy — Drug: bevacizumab 5mg/kg given by IV every 14 days. Other Name: Avastin
  Drug: cetuximab 400 mg/sqm initial dose, then 250 mg/sqm once weekly thereafter. Other Name: Erbitux
  Drug: oxaliplatin 8 5 mg/sqm by IV, day1. Component of mFOLFOX6.
  Drug: irinotecan 180 mg/sqm by IV, day1.Component of FOLFORI.
  Drug: calcium Folinate 400 mg/sqm by IV, day1.Component of mFOLFOX6 or FOLFORI.
  Drug: 5-fluorouracil 400 mg/sqm, day1,followed by 2400 mg/sqm iv infusion over 46~48 h.Component of mFOLFOX6 or FOLFORI.
  Arms: Investigator's Choice Chemotherapy

SUMMARY:
The main purpose of this study is to compare the clinical benefit, as measured by Progression-Free Survival (PFS), achieved by HX008 or Investigator's Choice Chemotherapy in participants with Microsatellite Instability High (MSI-H) or Mismatch Repair Deficient (dMMR) metastatic colorectal cancer (mCRC).

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the Informed Consent Form（ICF）, understand the study, be willing to follow and be able to complete all test procedures;
2. Male or female, age ≥ 18 years on the day of signing the informed consent form;
3. Subjects with colorectal cancer confirmed by histology are stage IV according to the 8th edition of the American Joint Committee on Cancer (AJCC) colorectal cancer tumor/node/metastasis (TNM) staging in 2017;
4. Confirmed MSI-H/dMMR status by the central laboratory;
5. No prior systemic treatment for metastatic colorectal cancer; subjects received neoadjuvant/adjuvant therapy with disease progression should be completed > 6 months prior to the neoadjuvant/adjuvant therapy were enrolled.
6. Has at least one measurable extracranial lesion (Lesions with the longest diameter ≥ 10mm, or lymph nodes with a short diameter ≥ 15mm) according to Response Evaluation Criteria in Solid Tumors Version 1.1(RECIST1.1), which has not been treated with local treatment(Lesions located in the area of previous radiation therapy can also optional if the progression is confirmed);
7. Eastern Cooperative Oncology Group (ECOG) of 0 or 1;
8. Estimated life expectancy of ≥12 weeks;
9. Has sufficient organ and bone marrow function((no blood transfusions allowed for 14 days prior to blood routine, no any cell growth factors or/and platelet-raising drugs) to meet the following laboratory examination standards:

   1. Absolute neutrophil count (ANC)≥1.5×10^9/L
   2. White blood cell count (WBC)≥3×10^9/L
   3. Platelet count (PLT)≥100×10^9/ L
   4. Hemoglobin (HGB)≥90 g/L
   5. Serum creatinine (Scr) ≤1.5×ULN
   6. Alanine aminotransferase (ALT) 、Aspartate aminotransferase (AST) ≤2.5× (upper limit of normal, ULN) . Patients with liver metastases require ALT and AST≤5×ULN,
   7. TBIL≤1.5×ULN
   8. International normalized ratio (INR) ≤ 2×ULN; or activated partial thromboplastin time (APTT)≤ 1.5×ULN;(except for patients on anticoagulant therapy);
10. Women of childbearing age must have a negative pregnancy test within 72 hours before the first dose of trial treatment. Reproductive men and women of childbearing age are willing to take adequate contraceptive measures (such as oral contraceptives, intrauterine contraceptives, sexual abstinence, or barrier contraceptives combined with spermicide) from signing the informed consent form to 12 months after the last administration of the trial drug;
11. The informed consent was voluntarily signed and the expected compliance was good.

Exclusion Criteria:

1. Prior systemic treatment for metastatic colorectal cancer (subjects who received neoadjuvant/adjuvant therapy with disease progression should be completed > 6 months prior to the neoadjuvant/adjuvant therapy were enrolled.)
2. Subjects diagnosed with any other malignancy within 5 years prior to randomization, except for malignancies with a low risk of metastasis and death (5-year survival rate > 90%), such as adequately basal cell or squamous cell skin cancer or carcinoma in situ of the cervix and other carcinomas in situ;
3. Had prior treatment with any anti-PD-1, anti-PD-L1, PD-L2, or CTLA-4 agent or any other drug targeting T cell co-stimulation or immune checkpoint pathway;
4. Has active autoimmune disease (except for psoriasis), that has required systemic treatment in the past 2 years((eg, corticosteroids or immunosuppressive drugs). Except for alternative therapies (eg, thyroxine, insulin or physiological corticosteroid replacement therapy for adrenal or pituitary insufficiency);
5. Need to receive systemic corticosteroids (dose equivalent to > 10 mg prednisone/day) or other immunosuppressive drugs within 14 days before enrollment or during the study period. Those under the following conditions are eligible:

   1. Locally external use or inhaled corticosteroids;
   2. short-term (≤ 7 days) use of glucocorticoids for the prevention or treatment of nonautoimmune allergic diseases;
6. Has had prior radiation therapy or has not recovered (≤ Grade 1 or at Baseline) from Adverse events(AEs) due to a previous radiation therapy;
7. Has received a significant surgery, open biopsy, or severe trauma within 4 weeks prior to randomization; Definition of major surgery: the minimum of 3 weeks of post-operative recovery time is required to undergo this study, any wound-related AE must be resolved prior to randomization;
8. Has severe infection within 4 weeks or active infection requiring IV infusion or oral administration of antibiotics within 2 weeks prior to randomization;
9. Has participated in other drug or device clinical trials within 4 weeks prior to randomization;
10. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis or found during screening;
11. Has uncontrolled ascites requiring repeated drainage, pleural effusion, or pericardial effusion;
12. Has incomplete intestinal obstruction, active gastrointestinal hemorrhage, or perforation;
13. Has a history or current interstitial pneumonia, or current non--infectious pneumonitis treatment with corticosteroids
14. Has uncontrolled cardiovascular disease, including but not limited to:

    1. heart failure greater than New York Heart Association (NYHA) class II
    2. unstable angina pectoris
    3. has myocardial infarction within 1 year
    4. supraventricular or ventricular arrhythmias with clinical significance poorly controlled without or despite clinical intervention;
15. Has uncontrolled systemic diseases, for instance, diabetes(Fasting Plasma Glucose ≥ 10 mmol/L or hypertension(systolic blood pressure ≥ 150 mmHg and / or diastolic blood pressure ≥ 100 mmHg);
16. Subjects with active tuberculosis;
17. History of human immunodeficiency virus infection, acquired or congenital immunodeficiency disease, organ transplantation, or stem cell transplantation;
18. Subjects with chronic hepatitis B or active hepatitis C. Except for Hepatitis B virus carriers or those with stable hepatitis B after drug treatment with DNA titer no higher than 500 IU/ml or copy number <2500 copies/ml, and cured hepatitis C patients (HCV RNA test negative);
19. Known to be allergic to macromolecular protein agents or monoclonal antibodies. Known to have a history of severe allergies to any of the chemotherapy drugs in the study ;
20. Alcohol dependence or drug abuse within the past 1 year;
21. Has received a live vaccine within 30 days prior to the first dose of trial treatment. Subjects are permitted to receive inactivated vaccines including those for seasonal influenza, intranasal influenza vaccines are not allowed;
22. Presence of other serious physical or mental illness or abnormal laboratory tests that may increase the risk of subjects in the study, or interfere with the study results, and the researchers believe that patients who are not suitable to participate in the trial for other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2022-12-20 (Estimated); Primary Completion 2026-01-19 (Estimated); Study Completion 2028-10-20 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) by Independent Review Committee(IRC) | 2 years
  PFS, defined as the time from randomization to the first documented disease progression per RECIST 1.1 assessed by IRC or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) by Investigators | 2 years
  PFS, defined as the time from randomization to the first documented disease progression per RECIST 1.1 assessed by investigators or death due to any cause, whichever occurs first.
Objective Response Rate (ORR) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) by IRC or investigators | 2 years
  ORR, defined as the percentage of subjects achieving complete response (CR) and partial response (PR).
Disease Control Rate (DCR) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) by IRC or investigators | 2 years
  DCR, defined as the proportion of subjects achieving CR, PR, and Stable disease(SD) after treatment.
Duration of Response (DOR) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) by IRC or investigators | 2 years
  DOR, defined as the duration from the initial recording of objective disease response to the first onset of tumor progression, or death of any cause.
Overall Survival (OS) | 2 years
  OS, defined as the duration from the start of treatment to death of any cause.
Immune Progression-free Survival (iPFS)-Experimental group per iRECIST assessed by IRC/investigators | 2 years
  iPFS, defined as the time from randomization to the first documented disease immune progression per iRECIST assessed by IRC/investigators or death due to any cause, whichever occurs first.
Immune Objective Response Rate (iORR)-Experimental group per iRECIST assessed by IRC/investigators | 2 years
  iORR, defined as the proportion of subjects with a best overall response (BOR) of immune complete response (iCR) or immune partial response (iPR) based on the immunotherapy Response Evaluation Criteria in Solid Tumors (iRECIST) by IRC/investigators.
Immune Disease Control Rate (iDCR) -Experimental group per iRECIST assessed by IRC/investigators | 2 years
  response, a partial response or stable disease according to immune Response Evaluation Criteria In Solid Tumors (iRECIST) criteria by IRC/investigators over the the total number of evaluable patients.
Immune Duration of Response (iDOR)-Experimental group per iRECIST assessed by IRC/investigators | 2 years
  iDOR, defined as the time from the date of the first immune response (iCR or iPR) to the date of immune confirmed progressive disease (iCPD) based on the immunotherapy Response Evaluation Criteria in Solid Tumors (iRECIST) by IRC/investigators.
Objective tumor response rate 2 (ORR2) (crossover phase) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) by IRC or investigators | 2 years
  ORR2, defined as proportion of subjects with best overall response of CR or PR, in progressors who continue to receive HX008 in crossover group.
Disease Control Rate 2 (DCR 2) (crossover phase) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) by IRC or investigators | 2 years
  DCR2, defined as the proportion of subjects achieving CR, PR, and SD after treatment who continue to receive HX008 in crossover group.
Duration of Response 2 (DOR2) (crossover phase) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) by IRC or investigators | 2 years
  DOR2, defined as the duration from the initial recording received HX008 in crossover group of objective disease response to the second onset of tumor progression, or death of any cause.
Progression-free Survival 2 (PFS2) (crossover phase) per Response Evaluation Criteria in Solid Tumors | 2 years
  PFS2, defined as duration of time until 2nd confirmed objective disease progression or death (or last documentation of being alive).
Immune Objective Response Rate 2 (iORR2) (crossover phase) per iRECIST assessed by IRC/investigators | 2 years
  iORR2, defined as the proportion of subjects with a best overall response (BOR) of immune complete response (iCR) or immune partial response (iPR) in progressors who continue to receive HX008 in crossover group based on the immunotherapy Response Evaluation Criteria in Solid Tumors (iRECIST) by IRC/investigators.
Immune Disease Control Rate 2 (iDCR2) (crossover phase) per iRECIST assessed by IRC/investigators | 2 years
  iDCR 2, defined as the percentage of patients whose best overall response is either a complete response, a partial response or stable disease who continue to receive HX008 in crossover group according to immune Response Evaluation Criteria In Solid Tumors (iRECIST) criteria by IRC/investigators over the the total number of evaluable patients.
Immune Duration of Response 2 (iDOR2) (crossover phase) per iRECIST assessed by IRC/investigators | 2 years
  iDOR2, defined as the time from the date of the first immune response (iCR or iPR) to the date of immune confirmed progressive disease (iCPD) who continue to receive HX008 in crossover group based on the immunotherapy Response Evaluation Criteria in Solid Tumors (iRECIST) by IRC/investigators.
Immune Progression-free Survival 2 (iPFS2) (crossover phase) per iRECIST assessed by IRC/investigators | 2 years
  iPFS2, defined as duration of time until 2nd confirmed objective disease progression or death (or last documentation of being alive) who continue to receive HX008 in crossover group based on the immunotherapy Response Evaluation Criteria in Solid Tumors (iRECIST) by IRC/investigators.
Adverse events | 2 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0, etc.

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Tianjin People's Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Xi'an

IPD SHARING:
Plan to Share IPD: No